CLINICAL TRIAL: NCT06725810
Title: A Prospective, Open-label, Randomized, Multicenter Study on the Rational Hemoglobin Target Value in Patients With Anemia of Non-dialysis Chronic Kidney Disease Treated With Enarodustat
Brief Title: Correction of Anemia With Enarodustat in Non-dialysis Dependent Chronic Kidney Disease
Acronym: CANNON
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-443
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Disease Associated Anemia
Keywords: HIF-PH inhibitor; anemia; chronic kidney disease; quality of Life; major adverse cardiovascular events; enarodustat
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — enarodustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- high-hemoglobin target group (Experimental): Patients are managed to achieve and maintain hemoglobin target of 13 g/dl over 96 weeks.
  Interventions: Drug: Enarodustat
- low-hemoglobin target group (Experimental): Patients are managed to achieve and maintain hemoglobin target of 11 g/dl over 96 weeks.
  Interventions: Drug: Enarodustat

INTERVENTIONS:
Drug: Enarodustat — Patients are administered with enarodustat with dosage adjusted according to hemoglobin levels to achieve and maintain hemoglobin target over 96 weeks.

SUMMARY:
The CANNON trial is a prospective, open-label, randomized, multicenter study designed to investigate rational hemoglobin target value in patients with anemia of non-dialysis chronic kidney disease treated with enarodustat. Eligible patients are randomly assigned 1:1 to the high-hemoglobin target group （hemoglobin of 13 g/dl）and low-hemoglobin target group （hemoglobin of 11 g/dl）and administered with enarodustat to achieve and maintain target hemoglobin over 96 weeks. The first primary endpoint was the difference of mean change in 36-Item Short Form Health Survey at week 24. The second primary endpoint was safety endpoints included time to major adverse cardiovascular + event (MACE+; all-cause mortality, myocardial infarction, stroke, and congestive heart failure requiring hospitalization) during 96 weeks.

DETAILED DESCRIPTION:
This study is a prospective, open-label, randomized controlled, multicenter investigation conducted among adult patients with ND-CKD anemia in China, with the aim of exploring the rational hemoglobin target value for the treatment of patients with ND-CKD anemia using enarodustat.

This study plans to enrol 1,670 patients with non-dialysis chronic kidney disease (ND-CKD) anemia. After screening, patients who meet the inclusion criteria and do not meet the exclusion criteria will be randomly assigned at a 1:1 ratio to: the low Hb target value group: with a Hb target value of 11 g/dL; the high Hb target value group: with a Hb target value of 13 g/dL. The initial dose of enarodustat tablets in both groups is 4 mg once daily. The dose will be adjusted in accordance with the instructions and the requirements of different Hb value groups.

The follow-up period will last for 96 weeks. The first primary endpoint was the difference of mean change in 36-Item Short Form Health Survey at week 24. The second primary endpoint was safety endpoints included time to major adverse cardiovascular + event (MACE+; all-cause mortality, myocardial infarction, stroke, and congestive heart failure requiring hospitalization) during 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years at the time of consent to participate;
2. Body weight ranged from 45 to 100 kg;
3. Diagnosed with CKD stages 2-5 (10 ≤ eGFR < 90 mL/min/1.73m2) and were not dialysis dependent;
4. Diagnosed with renal anemia:

1)Hemoglobin level of 6 - 10 g/dL for those who have not received ESA or HIF-PHI treatment within 6 weeks at screening; 2)Hemoglobin level of 8 - 12 g/dL for those who are currently receiving ESA (ESA dosage ≤ 10,000 IU/week) or HIF-PHI (roxadustat dosage≤ 100 mg TIW) at screening; 5. Serum ferritin > 100 μg/L or transferrin saturation > 20% at screening; 6. Voluntary participation in the trial and signing of the informed consent form.

Exclusion Criteria:

1. Uncontrolled hypertension identified as systolic blood pressure >160mmHg or diastolic blood pressure >100mmHg after 4 weeks of regular and adequate drug therapy prior to screening;
2. Uncontrolled proteinuria identified as UACR >3000mg/g or 24-hour urine protein >3.5g in non-diabetic patients and UACR of >5000mg/g or 24-hour urine protein >5.5g in diabetic patients;
3. Anemia due to other reasons except CKD including systemic hematological disorders (such as myelodysplastic syndrome, aplastic anemia, etc.), hemolytic anemia, hemorrhagic anemia or cancer-related anemia;
4. History of autoimmune diseases which could result in anemia such as systemic lupus erythematosus and ANCA vasculitis;
5. History of active bleeding within 4 weeks prior to screening;
6. History of serious thrombotic event such as a myocardial infarction, cerebral infarction, pulmonary embolism, unstable angina, or PCI or cardiac surgery within 6 months prior to screening;
7. Severe heart failure (NYHA class IV) at screening;
8. History of blood transfusion within 2 months prior to screening;
9. History of usage of immunosuppressants or other immune therapies within 6 months prior to screening;
10. Patients who are estimated to require dialysis, kidney transplantation, or major surgery within 6 months;
11. Severe liver and biliary system complications (AST or ALT >3 times the upper limit of normal, total bilirubin >2 times the upper limit of normal) at screening;
12. Receiving ESA combined with roxadustat treatment at screening;
13. History of proliferative retinopathy or diabetic retinopathy requiring ophthalmological treatment;
14. Severe hyperparathyroidism (iPTH ≥ 500 pg/mL);
15. Severe active infections (such as active tuberculosis, fungal infections, etc.);
16. Patients who are bedridden or have difficulty walking, or have a history of atrial fibrillation or deep vein thrombosis of the lower limbs;
17. History of active tumors;
18. Female patients who are pregnant or breastfeeding, or non-childbearing women who do not agree to effective contraception;
19. Patients with a history of severe drug allergies (such as anaphylactic shock), or known allergies to any of the active ingredients or excipients of enarodostat;
20. Patients who are currently participating in any other interventional clinical trial;
21. Other reasons determined by the investigator not suitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1670 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of quality of life | At week 24
  Mean change in 36-Item Short Form Health Survey
Effect on MACE+ events | During 96 weeks
  First occurence of major adverse cardiovascular + event (MACE+; all-cause mortality, myocardial infarction, stroke, and congestive heart failure requiring hospitalization) .

SECONDARY OUTCOMES:
Effect on blood transfusions | During 96 weeks
  Difference in the proportion of patients receiving blood transfusions between high- and low-hemoglobin target groups
Effect on thromboembolic events | During 96 weeks
  Diagnose thromboembolic events through clinical symptoms, laboratory tests, and auxiliary examinations. Compare the variance in the risk of thromboembolic events (excluding those in the cardiovascular system of the heart and brain) between high- and low-hemoglobin target groups
Effect on MACE events | During 96 weeks
  Diagnose MACE events （death from any cause, non-fatal myocardial infarction, non-fatal stroke）through clinical symptoms, laboratory tests, and auxiliary examinations. Dissimilarity in the risk of the first occurrence of MACE events between high- and low-hemoglobin target groups
Effect on cardiovascular death | During 96 weeks
  Discrepancy in the risk of cardiovascular death between high- and low-hemoglobin target groups
Effect on renal events | During 96 weeks
  Divergence in the incidence of renal events (defined as a reduction in eGFR by more than 50%, persistent dialysis for more than 3 months, or kidney transplantation) between high- and low-hemoglobin target groups
Effect on eGFR | At weeks 24, 48, 72, and 96
  Difference in the mean change of eGFR from baseline between high- and low-hemoglobin target groups

OTHER OUTCOMES:
Effect on the usage of iron agents | During 96 weeks
  Difference in the usage of iron agents between high- and low-hemoglobin target groups
Effect on the indices of iron metabolism | at weeks 12, 24, 48, 72, and 96
  Difference in the mean changes of ferritin, serum iron and transferrin saturation level from baseline between high- and low-hemoglobin target groups.
Difference of dosage of enarodostat | During 24 weeks
  Difference of mean dosage of enarodostat between high- and low-hemoglobin target groups
Evaluation of adverse drug events | during 96 weeks
  The variance of adverse drug events between high- and low-hemoglobin target groups

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqiang Ding, Principal Investigator — Fudan University
Locations (1):
- Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT06725810/Prot_SAP_ICF_000.pdf